CLINICAL TRIAL: NCT05621252
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Evaluation of PLN-74809 on Type 1 Collagen Deposition Using 68Ga-CBP8 PET/MRI Imaging in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Imaging Evaluation of PLN-74809 in Participants With IPF (PLN-74809)
Acronym: PLN-74809
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pliant Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLN-74809-IPF-205
Record Dates: First submitted 2022-11-02; First posted 2022-11-18 (Actual); Results first posted 2025-09-24 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: 2:1 randomization PLN-74809:placebo
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PLN-74809 (Experimental): 160 mg PLN-74809
  Interventions: Drug: PLN-74809
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PLN-74809 — 160 mg PLN-74809
  Arms: PLN-74809
Drug: Placebo — Matching placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2a, single -center, randomized, double-blind, placebo-controlled study to evaluate type 1 collagen deposition in the lungs following once-daily treatment with PLN-74809 for 12-weeks. This study is occurring at Massachusetts General Hospital.

DETAILED DESCRIPTION:
This is a Phase 2a, single-center, randomized, double-blinded, placebo-controlled study to evaluate type 1 collagen deposition in the lungs of participants with Idiopathic Pulmonary Fibrosis (IPF) following once-daily (QD) treatment with 160 mg PLN-74809 for 12 weeks. The study consists of an up to 28-day screening period, a 12-week treatment period, and a 2 week (±3 days) post treatment follow-up period.

Approximately 12 eligible participants will be randomized in a 2:1 ratio (160 mg PLN-74809 vs placebo; approximately 8 receiving PLN-74809 and 4 receiving placebo) on Day 1 (Visit 3). Randomization will be stratified by use of standard of care IPF therapy with pirfenidone or nintedanib. PET/MRI scans will be conducted at Baseline and at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Participants, aged 40 years or older
* Diagnosis of IPF, within 8 years prior to Screening
* FVC % predicted ≥45%; historical FVC for entry in the study is permitted if within 1 month of screening
* Diffusing capacity for carbon monoxide DLco (hemoglobin-adjusted) ≥30%; historical DLco for entry in the study is permitted if within 1 month of Screening
* Participants currently receiving treatment for IPF with nintedanib or pirfenidone are permitted, if on a stable dose for at least 3 months

Exclusion Criteria:

* Currently receiving or planning to initiate treatment for IPF (fibrosis) with agents not approved for that indication by the FDA
* Forced expiratory volume during the first seconds of the forced breath (FEV1)/FVC ratio <0.7 at Screening
* Clinical evidence of active infection, including but not limited to bronchitis, pneumonia, sinusitis that can affect FVC measurement or IPF progression
* Known acute IPF exacerbation or suspicion by the Investigator of such, within 6 months of Screening
* Smoking of any kind within 3 months of Screening

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2024-01-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sydney Montesi, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Montesi SB, Cosgrove GP, Turner SM, Zhou IY, Efthimiou N, Susnjar A, Catana C, Fromson C, Clark A, Decaris M, Barnes CN, Lefebvre EA, Caravan P. Dual alphavbeta6 and alphavbeta1 Inhibition over 12 Weeks Reduces Active Type I Collagen Deposition in Individuals with Idiopathic Pulmonary Fibrosis: A Phase 2, Double-Blind, Placebo-controlled Clinical Trial. Am J Respir Crit Care Med. 2025 Jul;211(7):1229-1240. doi: 10.1164/rccm.202410-1934OC. PMID 40153543

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PLN-74809 | Placebo
Started | 7 | 3
Completed | 7 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PLN-74809 | Placebo | Total
Number analyzed (Participants) | 7 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 3 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 3 | 9
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome
Description: Change from Baseline in top quartile whole lung PET standardized uptake value (SUV) following 12 weeks of treatment with PLN-74809. The whole lung SUV measures the intensity of the uptake of the radiotracer, 68GA-CBP8: peptide-based collagen binding probe 8 tagged with Gallium-68 radioisotope, in lung tissue. A negative change from baseline is a positive outcome and represents a decrease in the whole lung SUV corresponding to a decrease in collagen deposition in the lung. A positive change from baseline is a negative outcome and represents an increase in the whole lung SUV corresponding to an increase in collagen deposition in the lung.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Unitless
Arm/Group | PLN-74809 | Placebo
Number analyzed (Participants) | 7 | 3
Unitless | -0.0147 (0.10145) | 0.0740 (0.11839)

2. Secondary Outcome: Secondary Safety and Tolerability
Description: Safety and tolerability of PLN-74809 as measured by the incidence of adverse events.
Time Frame: From screening period (up to 28 days) to treatment period of 12 weeks, to 2 weeks after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | PLN-74809 | Placebo
Number analyzed (Participants) | 7 | 3
Participants | 6 | 1

3. Other Pre Specified Outcome: Exploratory 1
Description: Change from baseline in Forced vital capacity at 12 weeks.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PLN-74809 | Placebo
Number analyzed (Participants) | 7 | 3
mL | 21.4 (86.49) | -120.0 (84.85)

4. Other Pre Specified Outcome: Exploratory 2
Description: Change from baseline in Cough Severity Visual Analog Scale at 12 weeks. Cough severity is assessed on a 100-mm linear scale ranging from "no cough" (0mm) to "worst cough" (100mm). Higher score means worse outcome.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Mm
Arm/Group | PLN-74809 | Placebo
Number analyzed (Participants) | 7 | 3
Mm | -25.1 (29.11) | 40.3 (34.65)

ADVERSE EVENTS:
Time Frame: Bexotegrast Group: 84.9 [2.04] days; Placebo Group: 84.7 [0.58] days
Description: Adverse Events: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | PLN-74809 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 6/7 | 1/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PLN-74809 (N=7) | Placebo (N=3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lipase increased (Investigations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Per protocol, the data generated in this clinical study are the exclusive property of the Sponsor and are confidential. Any publication of the results of this study must be authorized by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/52/NCT05621252/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/52/NCT05621252/SAP_001.pdf